CLINICAL TRIAL: NCT01402089
Title: Cytochrom p450 3A4 and 1A2 Phenotyping for the Individualization of Treatment With Sunitinib or Erlotinib in Cancer Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Markus Joerger (Other)
Collaborators: University of Basel (Other)
Responsible Party: Sponsor-Investigator, Markus Joerger, MD-PhD-ClinPharm, Cantonal Hospital of St. Gallen
Organization: Cantonal Hospital of St. Gallen (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SG 327/10
Record Dates: First submitted 2011-07-20; First posted 2011-07-26 (Estimated); Last update posted 2016-02-02 (Estimated); Status verified 2016-01

CONDITIONS: Non Small-cell Lung Cancer; Renal-cell Cancer; Gastrointestinal Stroma Tumor
Keywords: phenotyping; cytochrome p450; erlotinib; sunitinib; lung cancer; renal-cell cancer; gastrointestinal stromal tumor
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Carcinoma, Renal Cell; Gastrointestinal Stromal Tumors; Lung Neoplasms | interventions — Sunitinib; Erlotinib Hydrochloride; Midazolam; Caffeine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Sunitinib — Patients with renal-cell cancer or GIST are receiving conventional treatment with sunitinib (50mg/day for 4 out of 6 weeks)
  Other Names: Sutent
Drug: Erlotinib — Patients with non small-cell lung cancer receive conventional treatment with erlotinib 150mg/day.
  Other Names: Tarceva
Drug: Midazolam — For phenotyping of CYP3A4, all patients receive one-time midazolam 2mg as a drinking solution at the start of study treatment.
  Other Names: Midazolam drinking solution
Drug: Caffeine — For phenotyping of CYP1A2, patients with non small-cell lung cancer receive additionally one-time caffeine 100mg as a tablet.
  Other Names: Coffeinum N 0.2g

SUMMARY:
It is well known that substantial interindividual variability of CYP3A4/1A2-phenotype activity is an important contributor to individual differences in the sensitivity to the frequently used tyrosine kinase inhibitors sunitinib and erlotinib. This study tests the potential for CYP-phenotyping to predict individual pharmacology and derive dosing algorithms for more tailored treatment of these drugs.

DETAILED DESCRIPTION:
Objectives:

The primary objective of this study is to show that the individual CYP3A4 and CYP1A2-phenotype as assessed by probe drugs predicts drug exposure to sunitinib and erlotinib. Secondary objectives of the study are to define the correlation between the individual CYP-phenotype and treatment-related toxicity, testing the feasibility of drug bioanalysis from patient's dry blood spots (DBS), build an integrated covariate model on sunitinib and erlotinib pharmacokinetics and define a dosing algorithm for both sunitinib and erlotinib based on the individual CYP-phenotype.

Study endpoints:

Primary endpoint:

• To show that individual drug clearance of sunitinib or erlotinib is significantly higher in patients with a high-activity CYP3A4/1A2-phenotype.

Secondary endpoints:

* To specify the correlation between the CYP-phenotype and treatment-related toxicity.
* To assess the feasibility of drug bioanalysis from patient's dry blood spots (DBS).
* To build an integrated covariate model of sunitinib and erlotinib pharmacokinetics to define the quantitative relationship between the CYP-phenotype activity and drug exposure.
* To define a dosing algorithm for both sunitinib and erlotinib based on the individual CYP-phenotype using data simulations on the previously defined population covariate model.

Trial Design:

Prospective, nonrandomized, pharmacological cohort study.

Main selection criteria

* Histologically or cytologically confirmed renal-cell cancer (sunitinib), gastrointestinal stromal tumor (sunitinib) or non small-cell lung cancer (erlotinib)
* Both early or advanced tumor stage
* Indication for the therapeutic use of either sunitinib or erlotinib
* Written informed consent and willing to undergo PK-sampling
* Adequate organ function
* No concurrent radiotherapy or systemic anticancer treatment with another drug

Trial Duration The present study is projected to start in June 2011, with the inclusion of a total of 60 patients (at least 25 patients for each sunitinib and erlotinib). The study is expected to finalize patient accrual in December 2013.

Statistical considerations The trial is designed to show a linear inverse relationship between the individual CYP-phenotype and total drug steady-state AUC (sunitinib plus SU12662 and erlotinib plus OSI-420, respectively), whereat CYP1A2 only accounts for the metabolism of erlotinib. With the inclusion of 60 patients, the study has a power of 90% to detect a relevant relationship between the CYP-phenotype activity and sunitinib/erlotinib steady-state AUC, with a regression coefficient of >0.4 for the H1-hypothesis (and accepting a regression coefficient of >0.1 for the H0-hypothesis) at the 5% significance level.

Trial Treatment Sunitinib: 50 mg p.o. daily for 4 out of 6 weeks, or 37.5 mg daily continuous until disease progression, unacceptable toxicity or withdrawal of informed consent.

Erlotinib: 150 mg p.o. daily until disease progression, unacceptable toxicity or withdrawal of informed consent.

Potential study outcome This study makes a significant contribution to global efforts for more individualized anticancer treatment. If successful, we will be able to make dosing recommendations for sunitinib and erlotinib based on a simple probe drug assay.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed renal-cell cancer or gastrointestinal stromal tumor (for sunitinib) or non small-cell lung cancer (for erlotinib)
* Both early or advanced tumor stage
* Indication for the therapeutic use of either sunitinib or erlotinib
* Written informed consent and willing to undergo PK-sampling
* Patients > 18 years of age
* ECOG performance status or ≤2
* Adequate laboratory parameters:

  i. Serum creatinine and serum bilirubin ≤ 1.5 X ULN ii. Serum ALT and AST ≤ 2.5 X ULN (or ≤ 5 in case of liver metastases) iii. Serum calcium ≤ 11,6 mg/dl (2.9 mmol/L)

Exclusion Criteria:

* Previous treatment with sunitinib or erlotinib
* Known hypersensitivity to trial drug or any compounds of the drug
* Concurrent radiotherapy
* Concurrent systemic anticancer treatment with the exception of bisphosphonates and bevacizumab in patients with non small-cell lung cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2012-01; Primary Completion 2015-07 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Steady-state partial area-under the plasma concentration-time curve over 24 hours (AUC24h) of sunitinib and erlotinib and CYP3A4/1A2-phenotype activity as defined in the protocol | 2 weeks
  Sunitinib or erlotinib area under the concentration-time curve during 24 hours at steady-state conditions, compared with the CYP3A4 or CYP1A2 phenotype activity as assessed by the two probe drugs midazolam (CYP3A4) and/or caffeine (CYP1A2)

SECONDARY OUTCOMES:
Sunitinib and Erlotinib-associated toxicity according to the CTC criteria (v.3.0) | 12 weeks (end of study)
Concentrations of Sunitinib, Erlotinib and probe drugs (Midazolam, Caffeine) in whole blood, sampled from patient's dried blood spots (DBS) | 12 weeks (end of study)
  Dried blood spots are a potential alternative to venous blood samples to assess drug exposure in cancer patients.

CONTACTS AND LOCATIONS:
Overall Officials: Markus Joerger, MD PhD, Study Chair — Cantonal Hospital of St. Gallen
Locations (1):
- Cantonal Hospital St.Gallen, Sankt Gallen, Switzerland